CLINICAL TRIAL: NCT06124833
Title: Building an Integrated Gut Microbiome Data Analysis Platform and Conducting Comparative Clinical Studies in Inflammatory Bowel Disease
Brief Title: Omics-driven Research on the Gut-Oral Microbiome, Metabolome, Lifestyle, and Clinical Integration in Korean Inflammatory Bowel Disease
Acronym: ORIGIN
Status: Recruiting | Type: Observational
Sponsor: Chang Kyun Lee (Other)
Collaborators: Kangbuk Samsung Hospital (Other); Chung-Ang University Hosptial, Chung-Ang University College of Medicine (Other); Inje University Haeundae Paik Hospital (Other); Yeungnam University Hospital (Other); Kyungpook National University Hospital (Other); Chonnam National University Hospital (Other); Wonkwang University Hospital (Other); Daejeon St. Mary's hospital (Other); Dankook University (Other); Kyung Hee University Hospital at Gangdong (Other); Inje University Ilsan Paik Hospital (Other); Hanyang University Guri Hospital (Other); Soon Chun Hyang University (Other); Chung-Ang University Gwangmyeong Hospital (Other); Keimyung University Dongsan Medical Center (Other)
Responsible Party: Sponsor-Investigator, Chang Kyun Lee, Professor, Kyunghee University Medical Center
Organization: Kyunghee University Medical Center (Other)
Other Study IDs: MB-IBD-01
Record Dates: First submitted 2023-10-25; First posted 2023-11-09 (Actual); Last update posted 2025-08-14 (Actual); Status verified 2025-08

CONDITIONS: Inflammatory Bowel Disease (IBD)
Keywords: Microbiota; Multiomics; Gut Microbiome; Oral Microbiome; Metabolome; Inflammatory Bowel Disease
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples With DNA — Plasma, tissue, stool, saliva, and DNA will be retained for central biobank
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Newly Diagnosed Cohort: Patients who have been diagnosed with inflammatory bowel disease (IBD, including Crohn's disease and ulcerative colitis) for the first time within the last 6 months prior to study enrollment.
- Disease Progression Cohort: Patients who were previously diagnosed with IBD and have been followed for over a year to understand disease progression and prognosis.
- Drug Cohort: Patients with IBD who, during their tracking observations, begin using biological agents and small molecule drugs for the first time.
- Familial IBD cohort: Cases where there are 2 or more diagnosed IBD patients among the patient's first-degree relatives (≥ 2 IBD-affected First Degree Relatives, FDR).
- Family Control Group: First-degree blood relatives of the patient who have never been diagnosed with IBD up to the point of study enrollment and who reside with the patient.

SUMMARY:
The inflammatory bowel disease (IBD) is a condition that afflects approximately 5 million people worldwide, with 1.4 million in the US and 2.2 million in Europe. By 2030, it is predicted that up to 1% of the entire Western population will have this disease. Notably, IBD encompasses conditions like Crohn's disease (CD) and Ulcerative colitis (UC). The emergence of this disease in non-Western countries is attributed to the rapid urbanization and industrialization which has led to the adoption of Westernized diets, an increase in the use of antibiotics early in life, and air pollution. These factors are suspected to induce changes in the gut microbiome, contributing to the rise of IBD. However, as an immune-mediated chronic intestinal disease, it is a multifactorial condition triggered by genetic mutations, gut microbial features, and environmental factors. Despite numerous studies, the exact causes remain insufficiently understood, emphasizing the importance of research and development to significantly benefit the health of the rapidly increasing patients. The study aims to construct a multi-omics analysis platform, including gut microbiome analysis, using biosamples collected from Korean patients with inflammatory bowel disease (IBD) and their families. Through this platform, comparative clinical research will be conducted to elucidate the pathophysiology of the disease and develop potential biomarkers.

DETAILED DESCRIPTION:
This study aims to construct a multi-omics analysis platform using biosamples collected from patients with inflammatory bowel diseases (IBD) and their families. Through this platform, comparative clinical research will be performed to elucidate the pathophysiology of the disease and develop potential biomarkers. The specific research objectives are as follows:

1. To identify clinical risk factors, genotype-genome variations, microbiome, and metabolomic markers that can predict high-risk groups prone to poor therapeutic outcomes and complications.
2. To elucidate differences in genotype, gut microbiome distribution, and metabolomics between non-responders to biological agents and small molecule drugs versus those with good therapeutic responses. Using this information, the aim is to develop multi-omics biomarkers that can predict responders and non-responders.
3. To develop a multi-omics biomarker-based algorithm that can prioritize the choice of various biological agents or small molecule drugs for individual patients.
4. To construct guidelines for precision treatment by identifying multi-omics markers associated with the onset of IBD, disease exacerbation, and complications and by clarifying the role of multi-omics in the pathophysiological mechanism.
5. Using familial IBD patients and family control groups, the study aims to elucidate environmental and genetic factors associated with the onset of IBD.
6. By comparing with the data of healthy intestines (non-blood-related disease control group), the role of gut microbiota in the pathogenesis of IBD and associated diseases in Koreans will be clarified.
7. By comparing with data from other target disease patients (e.g., AS, HIV), the role of gut microbiota in the onset of immune-mediated inflammatory diseases and associated conditions will be elucidated.
8. An integrated analysis of prior genomic data, current project genomic data (from the gut, oral-respiratory, skin, urogenital tracts), other domestic and international cohorts, and overseas genomic data will clarify regional and ethnic differences and roles of gut microbiota in the pathogenesis of IBD and associated diseases in Koreans.
9. To elucidate the interrelationship between human host genetic traits, microbiome, and environmental influences in the pathogenesis of IBD.

ELIGIBILITY:
Inclusion Criteria:

1. Korean patients with inflammatory bowel disease (including Crohn's disease and ulcerative colitis) aged between 13 and 85 years (at the time of participant consent).
2. First-degree blood relatives of the patient, aged between 13 and 85, who have never been diagnosed with IBD and reside with the patient (Family Control Group).
3. Participants who have received a detailed explanation about this clinical trial, fully understand it, have voluntarily decided to participate, and have given written consent to comply with the precautions.

Exclusion Criteria:

* For IBD patients

  1. Indeterminate colitis.
* For family control group

  1. Individuals with a history of using medications listed in Appendix 13 (Family Control Group Medication History) within a pre-specified period before the microbiome collection date.
  2. Individuals who have been vaccinated within the last month (4 weeks) prior to the microbiome collection date.
  3. Individuals who have applied topical antibiotics or topical steroids to the face, scalp, neck, or arms, forearms, hands within 24 hours prior to the microbiome collection date.
  4. Individuals who have used vaginal/external genital medications, including antifungals, within 24 hours prior to the microbiome collection date.
  5. Individuals with acute conditions (e.g., moderate or severe diseases with or without fever; however, sample collection can be postponed until the participant recovers).
  6. Individuals with chronic and clinically significant histories of liver, digestive, cardiovascular, renal, neurological, respiratory, endocrine, immune, hematological disorders, malignancies, psychiatric conditions, or a history of drug abuse.
  7. Individuals who have drastically changed their diet for rapid weight gain or loss within 4 weeks prior to the microbiome collection date.
  8. Individuals with gastrointestinal disorders that could impact microbiome analysis and are not currently medically managed or individuals under treatment for the following conditions: Inflammatory bowel diseases (e.g., Crohn's disease, ulcerative colitis), Irritable bowel syndrome (requiring drug therapy), Ulcers, acute or chronic pancreatitis, etc.
  9. Individuals requiring the use of incontinence diapers.
  10. Individuals with a positive urine pregnancy test, or who are pregnant or breastfeeding.
  11. Individuals suspected of having medical findings that may affect the sample collection at the time of microbiome sample collection.

Ages: 13 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Approximately 900 patients with inflammatory bowel disease (IBD) and about 200 first-degree relatives of the patients.
Sampling Method: Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2023-10-04 (Actual); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-08-01 (Estimated)

PRIMARY OUTCOMES:
Construction of a gut microbiome data platform by obtaining samples and clinical-related data from inflammatory bowel disease patients and control groups | 5 years
  Verify the input of clinical information for collected microbiome data. Confirm the number of collected microbiome biospecimens. Verify whether the collected microbiome biospecimens align with the research proposal objectives. Ensure the production and management of microbiome data collected.

SECONDARY OUTCOMES:
Production and measurement of multi-omics data | 5 years
  Host genomics, transcriptomics, metabolomics, proteomics, isolated bacterial strain

CONTACTS AND LOCATIONS:
Overall Officials: Chang Kyun Lee, MD, PhD, Principal Investigator — Kyunghee University Medical Center
Locations (1):
- Kyunghee University Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lloyd-Price J, Arze C, Ananthakrishnan AN, Schirmer M, Avila-Pacheco J, Poon TW, Andrews E, Ajami NJ, Bonham KS, Brislawn CJ, Casero D, Courtney H, Gonzalez A, Graeber TG, Hall AB, Lake K, Landers CJ, Mallick H, Plichta DR, Prasad M, Rahnavard G, Sauk J, Shungin D, Vazquez-Baeza Y, White RA 3rd; IBDMDB Investigators; Braun J, Denson LA, Jansson JK, Knight R, Kugathasan S, McGovern DPB, Petrosino JF, Stappenbeck TS, Winter HS, Clish CB, Franzosa EA, Vlamakis H, Xavier RJ, Huttenhower C. Multi-omics of the gut microbial ecosystem in inflammatory bowel diseases. Nature. 2019 May;569(7758):655-662. doi: 10.1038/s41586-019-1237-9. Epub 2019 May 29. PMID 31142855
- [Background] Kostic AD, Xavier RJ, Gevers D. The microbiome in inflammatory bowel disease: current status and the future ahead. Gastroenterology. 2014 May;146(6):1489-99. doi: 10.1053/j.gastro.2014.02.009. Epub 2014 Feb 19. PMID 24560869
- [Background] Integrative HMP (iHMP) Research Network Consortium. The Integrative Human Microbiome Project. Nature. 2019 May;569(7758):641-648. doi: 10.1038/s41586-019-1238-8. Epub 2019 May 29. PMID 31142853
- [Derived] Kim HS, Kim BH, Nam B, Oh SJ, Park SK, Lee SW, Lee JY, Jo S, Lee YA, Lee JY, Park DI, Kim TH, Lee CK. Oral-gut microbiome axis in a Korean cohort with inflammatory bowel disease and ankylosing spondylitis (INTEGRATE): a prospective and observational study protocol. BMJ Open. 2025 Aug 10;15(8):e092075. doi: 10.1136/bmjopen-2024-092075. PMID 40784769